CLINICAL TRIAL: NCT05839197
Title: A Single-arm, Exploratory Clinical Study of Hepatic Arterial Infusion Chemotherapy (HAIC) Combined With Apatinib and Camrelizumab in the Treatment of Unresectable Macrotrabecular-massive Hepatocellular Carcinoma
Brief Title: A Single-arm Clinical Study of HAIC Combined With Apatinib and Camrelizumab in the Treatment of Unresectable MTM HCC
Acronym: CCGLC-010
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wan-Guang Zhang (Other)
Responsible Party: Sponsor-Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202303126
Record Dates: First submitted 2023-04-15; First posted 2023-05-03 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Macrotrabecular Massive Hepatocellular Carcinoma
Keywords: HAIC; Camrelizumab; Apatinib
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC Combined With Apatinib and Camrelizumab (Experimental): All patients were treated with standard HAIC on the first day (D1). Immediately after the first HAIC, the liver function was reexamined. If the liver function was grade Child-Pugh A, Camrelizumab was given intravenously once every 3 weeks (D1) on the same day, 200mg/, once every 3 weeks (D1).
  Apatinib capsule was given orally to 250mg within half an hour after breakfast on the second day (D2) after the first HAIC. The drug was given continuously once a day and stopped on the same day of each HAIC.
  The combination of drugs for 3 weeks is a cycle.The treatment continued until the patient developed the disease or met the other criteria for terminating the study.
  Interventions: Procedure: HAIC; Drug: Camrelizumab plus Apatinib

INTERVENTIONS:
Procedure: HAIC — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 3 weeks.
  Other Names: hepatic arterial infusion chemotherapy of FOLFOX
Drug: Camrelizumab plus Apatinib — Apatinib(250 mg; p.o.; qd.); camrelizumab (200 mg; iv drip; q3w) If the liver function was grade Child-Pugh A, Camrelizumab was given intravenously once every 3 weeks (D1) on the same day, 200mg/, once every 3 weeks (D1).
  Apatinib capsule was given orally to 250mg within half an hour after breakfast on the second day (D2) after the first HAIC. The drug was given continuously once a day and stopped on the same day of each HAIC.

SUMMARY:
This is a single-arm, open, multicenter II phase clinical study to compare the efficacy and safety of HAIC combined with Apatinib and Camrelizumab in the treatment of unresectable middle-advanced MTM-HCC.

DETAILED DESCRIPTION:
Macrotrabecular-massive hepatocellular carcinoma (MTM-HCC) is a special pathological subtype of liver cancer, characterized by vascular invasion, early recurrence and poor survival. For unresectable MTM-HCC, there are currently no prospectively clinically validated treatment options. As a local interventional treatment, hepatic arterial infusion chemotherapy (HAIC) has shown better efficacy and safety than traditional transcatheter arterial chemoembolization (TACE) in the treatment of unresectable HCC. In addition, HAIC has been widely used as an alternative to sorafenib in advanced HCC in the eastern Asia. Studies have also shown that the combination of Apatinib and Camrelizumab has also shown encouraging results, and patients are well tolerated. Therefore, we designed HAIC combined with Apatinib and Camrelizumab for the exploratory study of unresectable MTM-HCC, in order to provide a safe, effective and tolerable option for patients with MTM-HCC, prolong their survival time and improve their quality of life.

Study population:

38 untreated patients with unresectable middle-advanced macrotrabecular-massive hepatocellular carcinoma

Treatment:

All patients were treated with standard HAIC (administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries) on the first day (D1).

Immediately after the first HAIC, the liver function was reexamined. If the liver function was grade Child-Pugh A, Camrelizumab was given intravenously once every 3 weeks (D1) on the same day, 200mg/, once every 3 weeks (D1).

Apatinib capsule was given orally to 250mg within half an hour after breakfast on the second day (D2) after the first HAIC. The drug was given continuously once a day and stopped on the same day of each HAIC.

The combination of drugs for 3 weeks is a cycle.The treatment continued until the patient developed the disease or met the other criteria for terminating the study.

Curative effect evaluation： The tumor condition was evaluated by imaging method at D28 (±7 days) after each HAIC, until the curative effect was evaluated as PD or unsuitable for further treatment. After 3 times of HAIC treatment, the tumor efficacy was evaluated every 8 weeks (±3 days) after the first HAIC treatment until disease progression (Response Evaluation Criteria In Solid Tumors（RECIST）1.1) or death (during treatment) or toxicity intolerable. The tumor treatment and survival status after disease progression were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Macrotrabecular Massive HCC diagnosed by histopathology or cytology according to the Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2022 Edition);
* Stage Ⅰa~Ⅱb and up-to-seven（tumor number +tumor size≥7) OR stage Ⅲa according to the Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2022 Edition);
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; expected survival ≥ 12 weeks;
* Child-Pugh liver function class A-B7
* Patients with newly diagnosed hepatocellular carcinoma who have not received any local or systemic treatment for hepatocellular carcinoma;
* At least one measurable lesion (according to RECIST1.1 standard); its diameter ≥ 1cm was accurately measured by magnetic resonance imaging (MRI) enhancement or computed tomography (CT) enhancement, and the target lesion had not received local treatment in the past (including not limited to hepatic arterial Infusion chemotherapy, radiofrequency ablation, argon-helium knife, radiotherapy, etc.);
* No serious organic diseases of heart, lung, brain and other organs;

Exclusion Criteria:

* Women who are pregnant (positive for pre-medication pregnancy test) or breastfeeding
* Participated in clinical trials of other antineoplastic drugs within 4 weeks before entering the group.
* Received any surgery or invasive treatment or operation (except venous catheterization, puncture and drainage, etc.) within 4 weeks before the start of the group;
* History of previous immune and targeted therapy for HCC;
* Patients who have previously received organ transplants or planned organ transplants;
* Significant clinical gastrointestinal bleeding or a potential risk of bleeding was identified by the investigator during the 30 days prior to study entry.
* Active or uncontrolled severe infection (≥ （Common Terminology Criteria for Adverse Events）CTCAE 2 grade infection);
* Suffered from other malignant tumors in the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical resection, or cervical carcinoma in situ;
* Any other disease, with clinically significant metabolic abnormalities, physical examination abnormalities or laboratory abnormalities, according to the researchers, there is reason to suspect that the patient has a disease or state that is not suitable for the use of research drugs (such as having seizures and requiring treatment), or will affect the interpretation of the results of the study, or put the patient at high risk;
* The researchers judged that patients have other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, and other serious diseases (including mental illness) that need to be combined with treatment. there are serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | After the first HAIC treatment, until the disease progresses or dies (during the treatment of the patient) or the toxicity is intolerable，through study completion, an average of 1 year
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including cases of complete remission (CR), partial remission (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of the first HAIC treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause.
Disease control rate (DCR) | From date of the first HAIC treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Percentage of confirmed cases including complete remission (CR), partial remission (PR) and disease stability (SD) among patients with evaluable efficacy
Total Survival time (OS) | Through study completion, an average of 2 year
  Refers to the date from the date of admission to the date of death of any cause
Incidence of adverse events and toxicities of Apatinib in combination with Camrelizumab | Until the last medication for 30 days (±7 days) or before the start of other anti-tumor therapy (whichever occurs first).
  Categorized according to NCI Common Toxicity Criteria version 5.0. Summarized in terms of type, severity (grade 1-5), and dose level in tabular format.

CONTACTS AND LOCATIONS:
Overall Officials: Wanguang Zhang, M.D.,Ph.D. Wanguang Zhang, M.D.,Ph.D., M.D.,Ph.D., Principal Investigator — Medical Ethics Committee of Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Hepatic Surgery Center, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China